CLINICAL TRIAL: NCT00810485
Title: A Phase 2B, Randomised, Double-blind, Placebo-controlled, Parallel Group, Dose-ranging, Multi-centre Study to Investigate the Efficacy, Safety and Tolerability of the mGluR5 Negative Allosteric Modulator ADX10059 in Patients With Gastroesophageal Reflux Disease (GERD) Who Are Partial Responders to Proton Pump Inhibitor (PPI) Treatment
Brief Title: ADX10059 as an add-on Therapy to Proton Pump Inhibitors (PPIs) in Patients With Gastroesophageal Reflux (GERD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Addex Pharma S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ADX10059-205; 2008-005105-18
Record Dates: First submitted 2008-12-17; First posted 2008-12-18 (Estimated); Last update posted 2012-07-16 (Estimated); Status verified 2012-07

CONDITIONS: Gastroesophageal Reflux
Keywords: Gastroesophageal reflux; Proton pump inhibitor; Heartburn; Regurgitation
MeSH Terms: conditions — Gastroesophageal Reflux; Heartburn

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- ADX10059 50 mg (Experimental): twice-daily
  Interventions: Drug: ADX10059
- ADX10059 100 mg (Experimental): twice-daily
  Interventions: Drug: ADX10059
- ADX10059 150 mg (Experimental): twice-daily
  Interventions: Drug: ADX10059
- ADX10059 Matching Placebo (Placebo Comparator): twice-daily
  Interventions: Drug: ADX10059 Matching Placebo

INTERVENTIONS:
Drug: ADX10059 — oral administration
  Arms: ADX10059 50 mg
Drug: ADX10059 — oral administration
  Arms: ADX10059 100 mg
Drug: ADX10059 — oral administration
  Arms: ADX10059 150 mg
Drug: ADX10059 Matching Placebo — oral administration
  Arms: ADX10059 Matching Placebo

SUMMARY:
The purpose of this study is to evaluate the effect of ADX10059 in patients with gastroesophageal reflux disease who are partial responders to proton pump inhibitors

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of typical GERD
* partial responder to a stable standard clinical symptoms control dose of PPI therapy
* body mass index ≤ 32 kg/m2

Exclusion Criteria:

* exclusively atypical symptoms of GERD
* symptoms that have been shown not to be associated with GERD
* erosive oesophagitis
* treated with a dose of PPI greater than the dose indicated for clinical symptom control of GERD
* hiatus hernia > 3 cm
* current diagnosis of co-existing psychiatric disease
* known clinical significant allergy or known hypersensitivity to drugs
* is pregnant or breast-feeding
* has received sodium valproate or topiramate within 30 days of Screening
* has a history of a significant medical condition that may affect the safety of the patient or preclude adequate participation in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2008-12; Primary Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Number of GERD symptom free days in week 4 of study medication treatment | 4 weeks

SECONDARY OUTCOMES:
GERD symptoms | 4 weeks
Sleep disturbance | 4 weeks
Use of antacid medications | 4 weeks
Global assessment of GERD | 4 weeks
Safety and tolerability assessments | 4 weeks

CONTACTS AND LOCATIONS:
Locations (40):
- United States (28):
  - Little Rock, Arizona
  - Tucson, Arizona
  - Anaheim, California
  - San Diego, California
  - Colorado Springs, Colorado
  - Jacksonville, Florida
  - Port Orange, Florida
  - Moline, Illinois
  - 54, Kansas City, Kansas
  - 62, Kansas City, Kansas
  - Jackson, Mississippi
  - Setauket, New York
  - Harrisburg, North Carolina
  - High Point, North Carolina
  - Huntersville, North Carolina
  - Raleigh, North Carolina
  - Winston-Salem, North Carolina
  - Fargo, North Dakota
  - Cleveland, Ohio
  - Oklahoma City, Oklahoma
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Germantown, Tennessee
  - 71, Nashville, Tennessee
  - 73, Nashville, Tennessee
  - Baytown, Texas
  - Houston, Texas
  - Waukesha, Wisconsin
- France (6):
  - Bordeaux
  - Colombes
  - Lyon
  - Nantes
  - Nice
  - Rouen
- Germany (4):
  - Dresden
  - Garmisch-Partenkirchen
  - Magdeburg
  - Munich
- Amsterdam, Netherlands
- Sankt Gallen, Switzerland